CLINICAL TRIAL: NCT01300013
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Safety and Efficacy of IV Infusion Treatment With Omecamtiv Mecarbil in Subjects With Left Ventricular Systolic Dysfunction Hospitalized for Acute Heart Failure
Brief Title: Study to Evaluate the Safety and Efficacy of IV Infusion Treatment With Omecamtiv Mecarbil in Subjects With Left Ventricular Systolic Dysfunction Hospitalized for Acute Heart Failure (ATOMIC-AHF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20100754
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: Intravenous; IV; Left Ventricular Systolic Dysfunction; Hospitalized; Acute heart failure; Heart failure; Left ventricular ejection fraction; pharmacokinetics; Pharmacodynamics; Dyspnea; hospitalization; In-patient; Omecamtiv mecarbil; Double-blind; Randomized; Placebo-controlled
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Dyspnea | interventions — omecamtiv mecarbil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Omecamtiv mecarbil (Experimental)
  Interventions: Drug: Omecamtiv mecarbil
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — 48-hour infusion of placebo
  Arms: Placebo
Drug: Omecamtiv mecarbil — 48-hour infusion of omecamtiv mecarbil; dose strength will depend on cohort assignment.
  Other Names: CK-1827452; AMG 423
  Arms: Omecamtiv mecarbil

SUMMARY:
The primary objective of the study is to evaluate the effect of 48 hours of intravenous (IV) omecamtiv mecarbil compared with placebo on dyspnea in subjects with left ventricular systolic dysfunction hospitalized for acute heart failure. This is a multicenter, randomized, double-blind, placebo-controlled study with 3 dose cohorts enrolled sequentially in order of ascending dose strength of omecamtiv mecarbil. In each cohort, subjects are randomized 1:1 to omecamtiv mecarbil or placebo.

DETAILED DESCRIPTION:
This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 85 years
* Hospitalized for worsening heart failure, within 24 hours of initiating IV loop diuretic
* Dyspnea due to heart failure, at rest or with minimal exertion
* History of left ventricular ejection fraction (LVEF) ≤ 40%
* Elevated brain natriuretic peptide (BNP) or N-terminal fragment BNP (NT-proBNP)

Exclusion Criteria:

* Receiving IV vasopressor (excluding low dopamine), inotropic or mechanical support
* Acute coronary syndrome (ACS)
* Within 30 days prior to enrollment: cardiac resynchronization therapy (CRT) or implantable cardioverter defibrillator (ICD) implantation, ACS, coronary revascularization, transient ischemic attack (TIA) or stroke, sustained ventricular arrhythmia, or major surgery
* Severe valvular stenosis, hypertrophic obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, or clinically significant congenital heart disease
* Estimated glomerular filtration rate (eGFR) < 20 mL/min/1.73m2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to evaluate the effect of 48 hours of intravenous (IV) omecamtiv mecarbil compared with placebo on dyspnea in subjects with left ventricular systolic dysfunction hospitalized for acute heart failure. | 48 hours

SECONDARY OUTCOMES:
To characterize pharmacokinetics of omecamtiv mecarbil including metabolites following IV infusion and to evaluate the relationship between omecamtiv mecarbil plasma concentration and echocardiographic parameters in subjects with AHF | 48 hours
To assess the safety and tolerability of 3 dose levels of IV omecamtiv mecarbil compared with placebo in subjects with left ventricular systolic dysfunction hospitalized for acute heart failure | 48 hours
To evaluate the effects of 48 hours treatment with IV omecamtiv mecarbil on additional measures of dyspnea, patient global assessment (PGA), change in NT-proBNP, incidence of worsening heart failure, and short term clinical outcomes | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (122):
- United States (41):
  - Research Site, Mobile, Alabama
  - Research Site, Inglewood, California
  - Research Site, La Jolla, California
  - Research Site, San Francisco, California
  - Research Site, Danbury, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Atlantis, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Novi, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Newark, New Jersey
  - Research Site, Cortlandt Manor, New York
  - Research Site, Roslyn, New York
  - Research Site, The Bronx, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Fairfield, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Murray, Utah
- Australia (5):
  - Research Site, Darlinghurst, New South Wales
  - Research Site, Woolloongabba, Queensland
  - Research Site, Bedford Park, South Australia
  - Research Site, Prahran, Victoria
  - Research Site, Richmond, Victoria
- Belgium (4):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Ghent
  - Research Site, Roeselare
- Bulgaria (7):
  - Research Site, Blagoevgrad
  - Research Site, Kazanlak
  - Research Site, Pazardzhik
  - Research Site, Plovdiv
  - Research Site, Sandanski
  - Research Site, Smolyan
  - Research Site, Sofia
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, QuÃ©bec, Quebec
  - Research Site, Sherbrooke, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Finland (2):
  - Research Site, Helsinki
  - Research Site, Turku
- France (6):
  - Research Site, Caen
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (12):
  - Research Site, Bad Nauheim
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Frankfurt
  - Research Site, Greifswald
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Homburg
  - Research Site, Langen
  - Research Site, Regensburg
  - Research Site, Stuttgart
  - Research Site, WÃ¼rzburg
- Greece (4):
  - Research Site, Athens
  - Research Site, Haidari
  - Research Site, Heraklion
  - Research Site, Pátrai
- Hungary (3):
  - Research Site, Budapest
  - Research Site, Pécs
  - Research Site, Szolnok
- Italy (4):
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Pavia
  - Research Site, Udine
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Netherlands (3):
  - Research Site, Delft
  - Research Site, Deventer
  - Research Site, Utrecht
- Norway (2):
  - Research Site, Oslo
  - Research Site, Stavanger
- Poland (6):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Wroclaw
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, St.-Petrsburg
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Nitra
- United Kingdom (4):
  - Research Site, Bristol
  - Research Site, Cottingham
  - Research Site, Glasgow
  - Research Site, Harrow

REFERENCES:
- [Derived] Teerlink JR, Felker GM, McMurray JJV, Ponikowski P, Metra M, Filippatos GS, Ezekowitz JA, Dickstein K, Cleland JGF, Kim JB, Lei L, Knusel B, Wolff AA, Malik FI, Wasserman SM; ATOMIC-AHF Investigators. Acute Treatment With Omecamtiv Mecarbil to Increase Contractility in Acute Heart Failure: The ATOMIC-AHF Study. J Am Coll Cardiol. 2016 Mar 29;67(12):1444-1455. doi: 10.1016/j.jacc.2016.01.031. PMID 27012405
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com